CLINICAL TRIAL: NCT01977729
Title: Sequencing CBT for Child Anxiety: CBT Plus Sertraline Versus Switch to Sertraline
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1308012517
Record Dates: First submitted 2013-10-30; First posted 2013-11-07 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Anxiety Disorder of Adolescence
Keywords: anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT with SRT (Experimental): CBT (Cognitive Behavioral Therapy)+SRT (Sertraline) will be scheduled at weeks 9-12, 14, 16, 18, 20 with telephone visits at weeks 15, 17, and 19. The same therapist as in Phase I will deliver CBT in Phase II, which will occur in conjunction with the psychiatrist visits. Phase II CBT will emphasize continued therapist prescribed in-session and out-of-session exposure tasks (developed with patient) and continued patient cognitive-affective processing of exposure sessions with therapist, with no instruction on new skills or therapeutic strategies. Therapists will be encouraged to discuss clinical status with patients, psychiatrists, and PIs to allow for treatment integration (e.g., psychiatrist could increase the dose of SRT, or not, depending on whether the patient Is making sufficient progress in CBT).
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Switch to SRT alone (Experimental): Sertraline is a selective serotonin reuptake inhibitor. Sertraline is FDA approved for the treatment of major depressive disorder, obsessive compulsive disorder, posttraumatic stress disorder, panic disorder, social anxiety disorder, and premenstrual dysphoric disorder in adults. Sertraline is also approved for the treatment of obsessive compulsive disorder in children and adolescents. Pharmacotherapy visits will be scheduled at weeks 9-12, 14, 16, 18, 20 with phone visits at weeks 15, 17, and 19. The psychiatrist will meet for ~30 min. with the youth and parents. Efforts will be made to use the most effective and tolerated SRT dose.
  Interventions: Drug: Sertraline; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Sertraline — Medication will be administered daily using a "fixed-flexible strategy" beginning at 25mg, titrating to 200mg across 8 wks (i.e., wks 9-17). We expect patients' medication dose will be adjusted upward in 50 mg/day increments if clinician-rated CGI-S anxiety severity is 3 (mild) or greater. The dose will be held or adjusted downward if patients have few anxiety symptoms (CGI-S<3) or impairing Adverse Events. Patients will be maintained at 200mg per day during wks 18-20.
  Other Names: Zoloft; Lustral
  Arms: Switch to SRT alone
Behavioral: Cognitive Behavioral Therapy — Youth are given instructions in each session that they may stop whenever they want and they do not need to attempt the task unless they so desire. Therapists have been carefully and thoroughly trained in providing reassurance and/or crisis treatments if needed. Therapists also have been trained to contact one of the PIs immediately in the event of a crisis.
  Other Names: CBT

SUMMARY:
The purpose of this study is to determine whether cognitive behavioral therapy (CBT) in combination with sertraline (SRT) is more effective than SRT alone in treating children and adolescents with anxiety disorders (after an initial 8 weeks of CBT).

DETAILED DESCRIPTION:
This project proposes to conduct a pilot study to collect preliminary data on a 'personalized adaptive treatment' approach for children and adolescents with anxiety disorders. All youth patients in this two site study will first receive CBT and all then will be re-assessed at mid-treatment (8 sessions). Patients who show a partial response or no response following 8 sessions of CBT will be randomized to either a switch to SRT alone or CBT augmentation with SRT.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for a primary Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) anxiety disorder of generalized anxiety disorder (GAD), social phobia (SOP), and separation anxiety disorder (SAD) using the DSM-5 version of the Anxiety Disorders Interview Schedule -Child and Parent Versions (ADIS-C/P)
* receive a mean score of 4 or greater on the ADIS-C/P Clinician Rating Scale of Severity (CSR)
* cease all other psychosocial treatment upon consultation with the clinic staff and the service provider
* not currently using any psychotropic medication other than a stable dose of stimulant medication treatment for comorbid ADHD. Youth who are on a stable dose of stimulant medication (i.e., a minimum of six months at the same dose) will be included so as not to limit generalizability.
* be between 8 and 16 years old
* have a negative pregnancy test, if they are menstruating girls. If participating in Phase II of the project (i.e., sertraline [SRT] vs. CBT + SRT) and they are sexually active, they must be using an appropriate method of birth control. Of additional note is that it is an allowable possibility to include children who have coexisting psychiatric diagnoses of lesser severity than the three target disorders including attention deficit-hyperactivity disorder (ADHD) while receiving stable doses of stimulant, obsessive compulsive, post-traumatic stress, oppositional defiant, and conduct disorders.

Exclusion Criteria:

* meet for primary diagnosis of any DSM-5 disorder other than GAD, SOP, and SAD
* have any of the following disorders (e.g., primary, secondary, tertiary) - Pervasive Developmental Disorders, Mental Retardation, Selective Mutism, Organic Mental Disorders, Bipolar Disorder, Tourette's Disorder, Schizophrenia and Other Psychotic Disorders. Drug or alcohol abuse/dependence will also be exclusionary.
* report the presence of any active suicidal ideation or a past suicide attempt in the last 6 months. Adolescents with a history of non-lethal self-harm behaviors (e.g., cutting) will be allowed to enroll if they meet other criteria
* have an intellectual disability as reported by guardian. If IQ is questionable or has not been assessed, the Block Design and Vocabulary subtests of the Wechsler Intelligence Scale for Children (WISC-IV) will be administered. If the youth receives an IQ subtest score < 6 on either one of these two subtests of the WISC-IV, a full scale IQ score (FSIQ) will be obtained. Children with FSIQ < 80 will be excluded
* be a victim of past or present undisclosed abuse requiring investigation or ongoing supervision by the Connecticut Department of Children and Families.
* have an unstable medical condition or a medical condition that could be worsened by selective serotonin reuptake inhibitors (SSRIs) such as a bleeding disorder or an active seizure disorder
* be using concomitant non-psychiatric medications that could be unsafe for use with sertraline (anticoagulants, triptans for migraine treatment, dextromethorphan)
* have a history of nonresponse to two adequate trials of SSRIs or an adequate trial of CBT or have a history of intolerance or nonresponse to sertraline
* be girls who are pregnant or are sexually active and are not using an effective method of birth control.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendry K. Silverman, Ph.D, Principal Investigator — Yale University Child Study Center
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Only one participant was recruited, but never randomized.
Period: Overall Study
Arm/Group | All Participants
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Severity & Improvement Scales
Description: Youth outcome will be assessed on a global level using the Clinical Global Impression (CGI) Severity Scale, ranging from 1 (not at all) to 7 (among the most extremely ill patients). Higher ratings indicate greater anxiety symptom severity. The CGI Improvement Scale ranges from 1 (very much improved) to 7 (very much worse). Lower ratings indicate greater improvement on anxiety symptom severity. A CGI Improvement Scale rating of 1 or 2 indicates clinically meaningful improvements in anxiety symptom severity.
Time Frame: 20 weeks from enrollment
Population: Medication was never given, and tests were never done.
Groups:
- CBT With SRT: CBT (Cognitive Behavioral Therapy)+SRT (Sertraline) will be scheduled at weeks 9-12, 14, 16, 18, 20 with telephone visits at weeks 15, 17, and 19.
- Switch to SRT Alone: Sertraline: Medication will be administered daily using a "fixed-flexible strategy" beginning at 25mg, titrating to 200mg across 8 wks (i.e., wks 9-17). We expect patients' medication dose will be adjusted upward in 50 mg/day increments if clinician-rated CGI-S anxiety severity is 3 (mild) or greater.
Arm/Group | CBT With SRT | Switch to SRT Alone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Multidimensional Anxiety Scale for Children
Description: Multidimensional Anxiety Scale for Children (MASC-2; Self-report and Parent completed). Treatment outcome will be assessed on a specific symptom level from the youth's and parent's perspective using the MASC-2. The MASC-2 consists of 50 items across 5 factors: Separation Anxiety/Phobias, Generalized Anxiety Disorder, Social Anxiety, Obsessions & Compulsions, and Harm Avoidance. MASC T-scores less than 65 indicate the child is no longer in the clinical range of anxiety symptoms.
Time Frame: 20 weeks from enrollment
Population: Study was terminated before randomization.
Arm/Group | CBT With SRT | Switch to SRT Alone
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Positive and Negative Affect Scale for Children
Description: Positive and Negative Affect Scale for Children (PANAS-C). Negative affect (NA) will be assessed using the NA subscale on the PANAS-C. The 15 NA items (e.g., sad, miserable) on the 27-item PANAS-C are scored 1 (very slightly or not at all) to 5 (extremely). Higher scores in the NA subscale indicate higher levels of negative affect.
Time Frame: 20 weeks from enrollment
Population: No data collected.
Arm/Group | CBT With SRT | Switch to SRT Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No adverse event data was collected before study termination.
Arm/Group | CBT With SRT | Switch to SRT Alone
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes